CLINICAL TRIAL: NCT03470454
Title: Prevalence of Contrast Nephropathy in Type 2 Diabetes Patients With Microalbuminuria
Brief Title: Contrast Nephropathy in Type 2 Diabetes
Acronym: VCG4
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of internal medicine, Fayoum University
Other Study IDs: VCG 4
Record Dates: First submitted 2018-03-09; First posted 2018-03-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Kidney Function Affection Upon Exposure to Radiocontrast; Diabetes; Microalbuminuria
MeSH Terms: conditions — Diabetes Mellitus | interventions — Linagliptin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- diabetics on linagelptin: Diabetic patients were given linagelptin for blood glucose control
  Interventions: Drug: Linagliptin Oral Tablet
- diabetics on other DPP4 inhibitors: Diabetic pateints were given other DPP4 inhibitors eg: vlidagliptin for blood glucose control
  Interventions: Drug: Linagliptin Oral Tablet

INTERVENTIONS:
Drug: Linagliptin Oral Tablet — Linagliptin for blood glucose control

SUMMARY:
To study the effect of radiocontrast material on kidney functions in diabetics with microalbuminuria

DETAILED DESCRIPTION:
Study design:

This study will be an observational prospective cohort study.

Study population:

Diabetics undergoing any intervention using radiocontrast material for any medical indication in Fayoum universiy hospital will be selected. There will be two arms of the study,each arm will contain 20 patients first arm diabetics on linagelptin, second arm diabetics on other DPP4 inhibitors.

Data collection:

Patients will be subjected to; full clinical examination,waist hip ratio assessment,BMI assessment fasting blood glucose,Serum uric acid, urine ACR, eGFR will be done before and after the investigation.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics on DPP 4 inhibitor treatment

Exclusion Criteria:

* Diabetics on insulin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetics undergoing any intervention using radiocontrast material for any medical indication in Fayoum university hospital will be selected.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
affection of estimated glomerular filtration rate | Two months
  A significant decrease in estimated glomerular filtration rate (eGFR)

SECONDARY OUTCOMES:
change in serum uric acid | Two months
  A significant rise in serum uric acid

OTHER OUTCOMES:
Affection of albumin creatinine ratio | Two months
  A significant increase in albumin creatinine ratio in urine (ACR)

CONTACTS AND LOCATIONS:
Overall Officials: Usama A Sharafeldin, MD, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of medicine Fayoum univesity, Al Fayyum
  - Fayoum University, Al Fayyum

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fayed A, Hammad AA, Abdulazim DO, Hammad H, Amin M, Elhadidy S, Salem MM, ElAzim IMA, Zsom L, Csongradi E, Soliman KM, Sharaf El Din UA. Is the combination of linagliptin and allopurinol better prophylaxis against post-contrast acute kidney injury? A multicenter prospective randomized controlled study. Ren Fail. 2023 Dec;45(1):2194434. doi: 10.1080/0886022X.2023.2194434. PMID 36974638